CLINICAL TRIAL: NCT03597802
Title: Effectiveness of Exercise at Workplace for Manual Material Handling Workers
Brief Title: Exercise at Workplace for Manual Material Handling Workers
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Universidade Cidade de Sao Paulo (Other)
Responsible Party: Principal Investigator, Rosimeire Simprini Padula, Professor, Universidade Cidade de Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2.372.435
Record Dates: First submitted 2018-04-29; First posted 2018-07-24 (Actual); Last update posted 2019-04-17 (Actual); Status verified 2019-04

CONDITIONS: Ergonomics; Manual Material Handling; Occupational Health
Keywords: Ergonomics; Workplace; Exercise
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (No Intervention): The workers will be receive orientation about manual material handling, postural and low back care (lecture and guidance).
- Intervention group 1 (Active Comparator): The workers will be receive orientation about manual material handling, postural and low back care (lecture and guidance), and will perform exercise at workplace three times per week, during 15 minutes
  Interventions: Other: Exercise at workplace - Four times per week
- Intervention group 2 (Active Comparator): The workers will be receive orientation about manual material handling, postural and low back care (lecture and guidance) and and will perform exercise at workplace four times per week, during 15 minutes.
  Interventions: Other: Exercise at workplace - Three times per week

INTERVENTIONS:
Other: Exercise at workplace - Three times per week — The exercise at workplace will be occur during the workday during the rest breaks. The exercises perform are stretching, and using load.
  Arms: Intervention group 2
Other: Exercise at workplace - Four times per week — The exercise at workplace will be occur during the workday during the rest breaks. The exercises perform are stretching, and using load.
  Arms: Intervention group 1

SUMMARY:
This study aim to evaluate the effectiveness of exercise at workplace for manual material handling workers. This is a randomized control trial study by cluster with three parallel groups (n=200). Participants will be randomized in three groups: (1) control group - will be receive ergonomics orientation . (2) Intervention group - exercise at workplace four times per week, during 15 minutes; (3) Intervention group 2 - exercise at workplace three times per week, during 15 minutes.Outcomes: The outcome measure will be verified in three moments at baseline, in six and eleven months of the intervention. The primary outcome is pain, electromyography. Secondary outcome is palmar dynamometer, BMI, physical activity level.

DETAILED DESCRIPTION:
Objective: This study aim to evaluate the effectiveness of exercise at workplace for control and prevention nonspecific low back pain. Methods: This is a randomized control trial study by cluster with three parallel groups. The context of this study is a motorcycle parts company importer localized in several states (Piaui, Ceará e Maranhão). The company has 575 workers, being 240 manual material handling. All are men over 18 years old that perform goods shipment (each work develop one this tasks - stock, separation, conference and packaging).

The inclusion criterial are workers that perform manual material handling for at least six months and signing informed consent form. The exclusion criterial were sick leave. The workers will be included with low back pain or no low back pain (at baseline). All will be interviewed to obtain: weight, height, BMI, age, marital status, educational level, and actual function (stock, separation, conference and packaging sick leave (the last 12 months), musculoskeletal complains, medications, complementary exams, surgery and or fractures. Participants will be randomized in three groups: (1) control group - will be receive orientation about manual material handling, postural and low back care (lecture and guidance). The training will be instructions according Ergonomics standard (NR17) about transportation and load handling and exercise in workout. (2) Intervention group 1 - will receive the same instruction of the control group, and will perform exercise at workplace four times per week, during 15 minutes; (3) Intervention group 2 - will be receive the same instruction of the control group, and will perform exercise at workplace three times per week, during 15 minutes. Outcomes: The outcome measure will be verified in three moments at baseline, six and eleven months of the intervention. The primary outcome is pain, electromyography. Secondary outcome is palmar dynamometer, BMI, exercise workout.

Expected Results: The manual material handling workers will be better after intervention by exercise at workplace. The effectiveness of exercise for low back pain and no low back pain groups will be contribute to change the behavior in occupational context.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criterial are workers that perform manual material handling for at least six months and signing informed consent form.

Exclusion Criteria:

* The exclusion criterial were sick leave

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — It is more common to be performed by men due to handled load
Enrollment: 240 (Estimated)
Dates: Start 2018-07-25 (Actual); Primary Completion 2018-12-19 (Actual); Study Completion 2020-12-17 (Estimated)

PRIMARY OUTCOMES:
Change from Pain Intensity at 6 months | At baseline and after six months
  Likert scale (0-10 points)
Change from electromyographic signal at 6 months | At baseline and after six months
  RMS (root mean square error) signal and peak signal by Electromyographic (EMG)

SECONDARY OUTCOMES:
Change from palmar grip strength at 6 months | At baseline and six months
  Three measure palmar grip strength to use the mean by dynamometer
Change from body mass index at 6 months | At baseline and after six months
  The body mass index will be calculated on height divided by square weight
Change of behavior to exercise | At baseline and after six months
  Practice of exercise (practice - yes or no; number of times per week)

CONTACTS AND LOCATIONS:
Locations (1):
- Rosimeire Simprini Padula, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No